CLINICAL TRIAL: NCT03073239
Title: Amyotrophic Lateral Sclerosis: a New Paradigm
Acronym: ALSParadigm
Status: Completed | Type: Observational
Sponsor: Conde, Bebiana, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2016-03-26; First posted 2017-03-08 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Bulbar disfunction; Rik factors ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood to test als mutations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS epidemiological characterization: epidemiological characterization
  Interventions: Other: ALS patients epidemiological caracterization
- Genetic findings in ALS patients: genética characterization
  Interventions: Genetic: ALS patients genetic characterization

INTERVENTIONS:
Genetic: ALS patients genetic characterization — Genetic findings in ALS patients
  Groups: Genetic findings in ALS patients
Other: ALS patients epidemiological caracterization — Epidemiological characterization in ALS patients
  Groups: ALS epidemiological characterization

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a degenerative neuromuscular disease, progressing inexorably to respiratory failure, the by involvement of respiratory muscles, the commitment with most impact on the prognosis of ALS.

According to current knowledge, the clinical presentation of the disease is characterized by spinal or bulbar involvement, the latter being associated with a worse prognosis.

There are multiple factors described in the aetiology of ALS, as the successive damage the motor neuron, which can happen in high-impact athletes, or exposure to heavy metals. Genetic mutations are also described, being associated to a higher prevalence of ALS.

Data from retrospective studies with ALS populations reveal a prevalence of 4-8 cases per 100,000 persons. Research carried out in Trás-os-Montes e Alto Douro region (Northeast of Portugal) shows a high prevalence of ALS, with near 10 cases per 100,000 persons, with a recent increase in the bulbar involvement. The reasons for the high prevalence of ALS in this region are unknown.

DETAILED DESCRIPTION:
The objective of this research is to pursue potentially involved genetic mutations in this disease (new or previously described), in addition to carry out a epidemiological questionnaire including data on personal history, environmental and occupational exposure that might be underlying this high prevalence.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Amyotrophic Lateral Sclerosis sent to a medical consultation

Exclusion Criteria:

* Amyotrophic Lateral Sclerosis not confirmed
* Ages less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Amyotrophic Lateral Sclerosis sent to a medical consultation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Finding environmental risk factor | 2 years
  Apply epidemiogycal form to All ALS patients sentido to respiratory evaluation in 2 years.

SECONDARY OUTCOMES:
Regional prevalence | 1 year
  Identify All cases ALS in regional area ( in north of Portugal)
Finding a genetic marker | 2 years
  Scan all ALS patients to eventually finding new ALS genes

CONTACTS AND LOCATIONS:
Overall Officials: Bebiana Conde, MD, Principal Investigator — Centro Hospitalar Tras-os-Montes e Alto Douro
Locations (1):
- Centro Hospitalar Tras-os-Montes e Alto Douro, Vila Real, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Research results will be shared with the scientific community through the publication of 2 to 3 papers in medical journals, as well as through the participation in national and international conferences. Whenever requested by the participants, the individual data resulting from clinical examinations will be provided.